CLINICAL TRIAL: NCT06078436
Title: Pulmonary Artery Catheterization and Carvedilol Early Initiation in Cardiogenic SHOCK Caused by Heart Failure With Reduced Ejection Fraction
Brief Title: Pulmonary Artery Catheterization and Carvedilol Early Initiation in Cardiogenic SHOCK Due to HFrEF
Acronym: PACE-SHOCK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Min-Seok Kim (Other)
Responsible Party: Sponsor-Investigator, Min-Seok Kim, Clinical Associate Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC_2023_0794
Record Dates: First submitted 2023-09-20; First posted 2023-10-11 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Cardiogenic Shock
Keywords: Cardiogenic shock; Heart failure with reduced ejection fraction (HFrEF); Hemodynamic monitoring; Pulmonary artery catheter; Carvedilol
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Intervention Model Description: From the time of diagnosing cardiogenic shock (CS) caused by HFrEF within 12 hours, random allocation will be conducted. If assigned to the hemodynamic monitoring group with pulmonary artery catheter (PAC), the catheter will be inserted and hemodynamic parameters will be monitored until recovery from CS. The non-monitoring group will receive CS treatment without inserting a PAC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary artery catheter monitoring group (Experimental): Within 8 hours of random allocation, a pulmonary artery catheter will be inserted to monitor hemodynamic parameters.
  Interventions: Device: Pulmonary artery catheter
- No pulmonary artery catheter monitoring group (Active Comparator): After random allocation, a pulmonary artery catheter will not be inserted during cardiogenic shock management.
  Interventions: Device: Pulmonary artery catheter

INTERVENTIONS:
Device: Pulmonary artery catheter — Pulmonary artery catheter monitoring or not
  Other Names: Swan-Ganz catheter

SUMMARY:
This study aims to compare the impact of hemodynamic monitoring using pulmonary artery catheter (PAC) on survival and inotropic agent reduction in patients with cardiogenic shock caused by heart failure with reduced ejection fraction (HFrEF). The investigators also intend to compare the difference in long-term survival rates among patients who have recovered from cardiogenic shock due to HFrEF, based on the timing of initiation of beta-blocker treatment.

DETAILED DESCRIPTION:
Cardiogenic shock is one of the most common causes of shock patients admitted to the Cardiac Intensive Care Unit (CICU). Despite advances in treatment, the mortality rate of cardiogenic shock remains high, up to 50%, and improving survival is crucial through the use of inotropic agents, vasopressors, or mechanical circulatory support devices to improve hemodynamic parameters. Previous meta-analyses of retrospective studies have shown the usefulness of pulmonary artery catheter monitoring, especially in patients with cardiogenic shock due to heart failure. However, there is a lack of prospective studies regarding specific monitoring indicators and treatment goals. This study aims to compare the impact of hemodynamic monitoring through pulmonary artery catheter on survival and inotropic agent reduction in patients with cardiogenic shock caused by heart failure with reduced ejection fraction.

In the PAC non-monitoring group, various assessments such as physical examination, echocardiographic findings, serum lactate levels, chest x-ray, and laboratory test results are utilized. If there are signs of volume overload, diuretics or hemodialysis may be applied to achieve for volume reduction. The dosage of diuretics and the timing of hemodialysis are at the discretion of the attending physician. The target of a mean arterial pressure (MAP) is 65mmHg or higher. If the MAP falls below 65mmHg, increasing vasopressor or inotropes should be considered. If the MAP target is not achieved with medical therapy or if serum lactate levels increase by 3 mmol/L or more compared to the lowest value within 24 hours, mechanical circulatory support (MCS) is considered. The specific dosage of vasopressors/inotropes and the timing of MCS application are at the dscretion of the attending physician.

The PAC monitoring group, in addition to those used in the PAC non-monitoring group, treats patients using indicators measured by PAC. The targets include a right atrial pressure (RAP) or central venous pressure (CVP) of 8mmHg or lower and pulmonary capillary wedge pressure (PCWP) of 15mmHg or lower. Whan RAP or CVP exceeds 8mmHg, or PCWP exceeds 15mmHg, employing diuretics or hemodialysis should be considered for volume reduction. The dosage of diuretics and the timing of hemodialysis are at the discretion of the attending physician. The target of a mean arterial pressure (MAP) is 65mmHg or higher. If the MAP falls below 65mmHg, increasing vasopressor or inotropes should be considered. If the MAP target is not achieved with medical therapy or if serum lactate levels increase by 3 mmol/L or more compared to the lowest value within 24 hours, mechanical circulatory support (MCS) is considered. The specific dosage of vasopressors/inotropes and the timing of MCS application are at the dscretion of the attending physician.

Additionally, the beta-blocker Carvedilol is known to reduce mortality and readmission rates in heart failure patients based on large-scale clinical trials and is widely prescribed as a standard treatment. However, the evidence for the appropriate timing of Carvedilol initiation and objective indicators of hemodynamic stability beyond the point of discharge is currently insufficient, relying solely on the clinical judgment and experience of the treating physician. Through subgroup analysis, the investigators intend to compare the difference in long-term survival rates among patients who have recovered from cardiogenic shock due to heart failure with reduced ejection fraction, based on the timing of iniation of beta-blocker treatment. The early administration of Carvedilol is defined as initiating treatment within 24 to 48 hours after discontinuing vasopressor/inotropic agents or mechanical circulatory support in stable condition following cardiogenic shock. The conservative administration of Carvedilol is defined as initiating treatment at least 48 hours after discontinuing vasopressors/inotropic agents or mechanical circulatory support in stable condition following cardiogenic shock.

Also, lung B-line will be measure along with PAC measured hemodynamic parameters using lung ultrasound at eight regions of the thorax in patients with PAC monitoring. Number of B-line in a total and each region, positive region which is defined as having three or more number of B-line will be recorded. Acquired images will be adjudicated by two investigators who are blinded to the clinical information of the subject.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 19 and above ( no age limit for elderly )
* Patients with cardiogenic shock requiring intensive care monitoring in ICU
* Patients eligible for oral medication administration
* Patients who have provided research participation consent through a written informed consent form

Exclusion Criteria:

* Unwilling or unable to obtain informed consent by the participant or substitute decision maker
* Patients with mechanical circulatory support at the time of screening
* Patients with acute coronary syndrome
* Patients with severe valvular heart disease requiring emergent percutaneous procedures or surgery
* Known hypersensitivity to beta-blockers
* Patients with a history of bronchospasm or asthma
* Patients with bradycardia or second or third-degree atrioventricular block
* Patients with sick sinus syndrome, including sinoatrial block
* Patients with untreated pheochromocytoma
* Patients currently undergoing de-sensitization therapy
* Patients who are currently pregnant, postpartum period within 30 days or breast-feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
30-day all-cause mortality | From date of randomization until the date of death from any cause, assessed up to 30 days
  All-cause mortality

SECONDARY OUTCOMES:
All-cause mortality | From date of randomization until the date of death from any cause, assessed up to 3 months
  All-cause of death
Cardiovascular mortality | From date of randomization until the date of death from any cause, assessed up to 3 months
  Cardiovascular death
Timing of discontinuation of inotropic or vasopressor agents | From date of randomization until the date of discharge or assessed up to 90 days
  Days from randomization to discontinuation of inotropes/vasopressor
The rate of Carvedilol intake on the 3 months | 3 months from date of randomization
  The rate of Carvedilol intake
The target-dose achievement rate of Carvedilol on the 3 months | 3 months from date of randomization
  Target dose : 50mg/day
3-month follow-up echocardiography parameters | 3 months from date of randomization
  LVEF(left ventricular ejection fraction)
Complications related with pulmonary artery catheter | During hospitalization period, up to 30 days
  Any complications related with pulmonary artery catheter
Hospitalization due to heart failure | 3 months from date of randomization
  Unplanned hospitalization due to heart failure
The composite outcome of cardoivascular death and heart failure hospitalization | 3 months from date of randomization
  The composite outcome of cardiovascular death and hospitalization due to heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Min-Seok Kim, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No